CLINICAL TRIAL: NCT01068483
Title: A Phase IA, Multicenter, Open-label Dose Escalation Study of BKM120, Administered Orally in Adult Patients With Advanced Solid Malignancies
Brief Title: Safety of BKM120 Monotherapy in Advanced Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120X2101; 2008-002652-17 (EudraCT Number)
Record Dates: First submitted 2010-02-11; First posted 2010-02-15 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2013-04

CONDITIONS: Breast Cancer; Colon Cancer; Ovarian Cancer; Endometrium Cancer
Keywords: Advanced solid tumors; Breast Cancer; Colon Cancer; Ovarian Cancer; Endometrium cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 (Experimental): Dose escalation followed by dose expansion
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120

SUMMARY:
This is a first-in-man, phase I clinical research study with BKM120, a potent and highly specific oral pan-class I phosphatidylinositol-3-kinase (PI3K) inhibitor. The study consists of a dose escalation part followed by a MTD expansion part.

Once the MTD has been defined, the MTD expansion part will be opened for enrollment.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Histologically-confirmed advanced solid tumors
* Progressive, recurrent unresectable disease
* World Health Organization (WHO) Performance status ≤ 2
* No history of primary brain tumor or brain metastases

MTD Expansion part:

* Histologically-confirmed advanced solid tumors
* Progressive, recurrent unresectable disease
* World Health Organization (WHO) Performance status ≤ 2
* No history of primary brain tumor; no brain metastases unless asymptomatic and clinically stable for ≥ 3 months
* Patients with genetic or molecular alteration of the PI3K pathway

Exclusion Criteria:

* Prior treatment with a PI3K inhibitor
* History of or active major depressive episode, bipolar disorder, schizophrenia, or history of suicidal attempt or ideation
* No clinically manifest diabetes mellitus (treated and/or with clinical signs)
* No acute or chronic renal disease
* No acute or chronic liver disease
* No acute or chronic pancreatitis
* No unresolved diarrhea
* No impaired cardiac function or clinically significant cardiac diseases such as ventricular arrhythmia, congestive heart failure, uncontrolled hypertension
* No acute myocardial infarction or unstable angina pectoris within the past 3 months
* Not pregnant or nursing and fertile patients must use barrier contraceptives

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BKM120 | throughout the study

SECONDARY OUTCOMES:
Safety and tolerability of BKM120 | throughout the study
Pharmacokinetics of BKM120 | throughout the study
Changes in tumor metabolic activity | throughout the study
Pharmacodynamics of BKM120 | throughout the study
Clinical tumor response in patients with tumors that show PI3K pathway activation | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Sarah Cannon Research Institute Dept.ofSarahCannonCancerCtr(4), Nashville, Tennessee, United States
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- See also: Results for CBKM120X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7084